CLINICAL TRIAL: NCT06435273
Title: A Randomised, Double-blind, Parallel Group, Placebo Controlled, 4-Week, Phase II Study to Evaluate the Effect of AZD4604 on Airway Inflammation and Biomarkers in Adults With Asthma
Brief Title: Phase II Study to Evaluate the Effect of AZD4604 on Airway Inflammation and Biomarkers in Adults With Asthma
Acronym: ARTEMISIA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D8210C00005; 2023-510291-32-00 (Registry Identifier: CTIS)
Record Dates: First submitted 2024-05-24; First posted 2024-05-30 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Asthma
Keywords: Asthma, Mechanistic Study, Bronchoscopy
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AZD4604 (Experimental): AZD4604
  Interventions: Drug: AZD4604
- Placebo to AZD4604 (Placebo Comparator): Placebo to AZD4604
  Interventions: Drug: Placebo to AZD4604

INTERVENTIONS:
Drug: AZD4604 — Janus kinase 1 (JAK1) inhibitor
  Other Names: Londamocitinib
  Arms: AZD4604
Drug: Placebo to AZD4604 — Placebo to AZD4604
  Arms: Placebo to AZD4604

SUMMARY:
The purpose of this study is to investigate the effect on airway inflammation and JAK1-associated signalling pathways of AZD4604 compared with placebo in participants with moderate-to-severe asthma.

Study details include:

* The study duration for each participant will be approximately 10 weeks.
* The duration of IMP administration will be approximately 4 weeks.

DETAILED DESCRIPTION:
This is a multicentre, randomised, placebo-controlled, double-blind study to investigate the effect on airway inflammation and JAK1-associated signalling pathways of AZD4604, administered over a 4-week treatment period to adult patients with moderate-to-severe asthma. The study will recruit patients receiving treatment with medium-to-high dose inhaled corticosteroid-long-acting beta-agonist (ICS-LABA) at screening and having a history of at least one severe asthma exacerbation within the year prior to Visit 1 or have an Asthma control questionnaire-6 (ACQ-6) score ≥ 1.5 at Visit 1. Enrolled participants will be randomised into the study to either AZD4604 or placebo. Participants discontinuing the study before the completion of Visit 6a (including the second bronchoscopy) will be replaced. Participants will be randomised using an interactive response technology/randomisation and trial supply management system at a ratio of 2:1 to AZD4604 or placebo, respectively. Randomisation will be stratified based on fractional exhaled nitric oxide (FeNO) levels to ensure a similar proportion of participants with FeNO above and below 25 parts per billion (ppb) in the 2 treatment arms. The study will be conducted at approximately 28 sites in approximately 6 countries.

ELIGIBILITY:
Inclusion Criteria:

* Documented physician-diagnosed asthma ≥ 12 months prior to screening (Visit 1).
* Participants treated with medium-to-high dose ICS in combination with LABA at a stable dose for at least 2 months prior to Visit 1 (the ICS can be contained within an ICS-LABA fixed dose combination product or as separate inhaled products regularly taken together). Treatment with additional asthma controller therapies (eg, long-acting muscarinic antagonist, leukotriene receptor antagonist) at a stable dose ≥ 2 months prior to Visit 1 is allowed. Treatment with maintenance systemic corticosteroids (oral or injectable) is not allowed.
* A documented history of ≥ 1 severe asthma exacerbation within 1 year prior to Visit 1 or ACQ-6 ≥ 1.5 at Visit 1. A severe asthma exacerbation is defined as a worsening of asthma that leads to an inpatient hospitalisation (defined as admission to an inpatient facility and/or evaluation and treatment in a healthcare facility for ≥ 24 hours) due to asthma.
* Morning pre-BD FEV1 ≥ 60% predicted at Visit 1.
* Able to perform acceptable lung function testing for FEV1 according to American Thoracic Society/ European Respiratory Society (ATS/ERS) 2019 acceptability criteria.
* Able and willing to undertake bronchoscopy. There should be no absolute contra-indications to bronchoscopy as outlined in the bronchoscopy manual.
* Documented evidence of asthma in the 5 years up to or including Visit 1.
* Able and willing to comply with the requirements of the protocol including ability to read, write, be fluent in the translated language of all participant-facing questionnaires used at the study site, and use electronic devices, eg, electronic patient reported outcomes (ePRO) device and spirometer.
* Body weight ≥ 40 kg and body mass index < 35 kg/m2.
* All females must have a negative serum pregnancy test result at Visit 1.
* Females not of childbearing potential are defined as females who are either permanently sterilised (hysterectomy, bilateral oophorectomy, or bilateral salpingectomy), or who are postmenopausal.
* All FOCBP who are sexually active with a non-sterilised male partner must agree to use one highly effective method of birth control.

Highly effective birth control methods include:

* Non-hormonalTotal sexual abstinence provided it is the usual lifestyle of the participant (defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatments)
* A vasectomised partner (with confirmed absence of sperm in semen)
* Bilateral tubal occlusion (caveat: failure rate >1%)
* Intrauterine device (copper)Hormonal
* Levonorgestrel intrauterine system
* Medroxyprogesterone injections
* Combined oral or transdermal contraceptives (ethinyl estradiol plus progestin) o Intravaginal device (eg, EE and etonogestrel)

The following are not acceptable methods of contraception:

* Periodic abstinence (calendar, symptothermal, post-ovulation methods)
* Withdrawal (coitus interruptus)
* Spermicides only
* Lactational amenorrhoea
* Female condom and male condom should not be used together

Exclusion Criteria:

* A severe asthma exacerbation within 8 weeks prior to Visit 1.
* History of herpes zoster reactivation (shingles).
* Clinically important pulmonary disease other than asthma, eg, active lung infection, chronic obstructive pulmonary disease (COPD), bronchiectasis, pulmonary fibrosis, cystic fibrosis, hypoventilation syndrome associated with obesity, lung cancer, history or planned lung lobectomy, alpha-1 anti-trypsin deficiency, primary ciliary dyskinesia, Churg-Strauss syndrome, allergic bronchopulmonary aspergillosis, and hyper-eosinophilic syndrome.
* Any disorder, including, but not limited to, cardiovascular, gastrointestinal, hepatic, renal, neurological, musculoskeletal, infectious, endocrine, metabolic, haematological, psychiatric, or major physical impairment that is not stable in the opinion of the investigator.
* Any clinically significant cardiac or cerebrovascular disease.
* History of venous thromboembolism.
* Participants with a recent history of, or who have a positive test for, infective hepatitis or unexplained jaundice, or participants who have been treated for hepatitis B, hepatitis C, or human immunodeficiency virus (HIV). Positivity for hepatitis B virus (HBV) surface antigen is a reason for exclusion.
* Current or prior history of alcohol or drug abuse (including marijuana), as judged by the investigator. Positive drug screening result that cannot be justified by participant's medical history and its relevant treatment (over-the-counter product or a valid prescription), or history of or current alcohol or drug abuse (including marijuana and marijuana-containing valid prescriptions), as judged by the investigator.
* History of malignancy other than superficial basal cell carcinoma.
* Treatment with systemic corticosteroid (short-term or maintenance) use within 8 weeks (oral) or 12 weeks (intramuscular) before Visit 1.
* Any immunosuppressive therapy (including hydroxychloroquine, methotrexate, cyclosporine, and tacrolimus) within 12 weeks prior to Visit 1.
* Treatment with marketed biologics including benralizumab, mepolizumab, reslizumab, omalizumab, dupilumab, and tezepelumab within 6 months or 5 half-lives of Visit 1, whichever is longer.
* Inhaled corticosteroid plus fast-acting β2 agonist as a rescue medication (eg, Symbicort, Fostair, or Airsupra Maintenance and Reliever Treatment) is not allowed 30 days prior to Visit 1, during screening, run-in and baseline periods, throughout the treatment period, and preferably until 1 week after the last administration of the IMP.
* Live, attenuated, or mRNA vaccines within 4 weeks of Visit 1.
* Immunoglobulin therapy or blood products within 4 weeks of Visit 1.
* Any immunotherapy within 6 months of Visit 1, except for stable maintenance dose allergen-specific immunotherapy started at least 4 weeks prior to Visit 1 and expected to continue through to the end of the follow-up period.
* Anticoagulants (including vitamin K antagonists and Factor Xa inhibitors). Antiplatelet agents are allowable if in the opinion of the investigator they can be safely withheld for 7 days prior to the procedure.
* Any history of bronchial thermoplasty
* Participants with a known hypersensitivity to AZD4604 or any of the excipients of the product.
* Abnormal findings identified on physical examination, ECG, or laboratory testing include, but not limited to: Alanine aminotransferase/transaminase (ALT) or aspartate aminotransferase/transaminase AST ≥ 1.5 × upper limit of normal (ULN), Total bilirubin (TBL) ≥ ULN (unless due to known Gilbert's disease), Evidence of chronic liver disease, International Normalised Ratio (INR) > 1.5, Platelet count < 150,000 per microliter, Abnormal vital signs, after 5 minutes of supine or sitting rest (confirmed by 1 controlled measurement), defined as any of the following: Systolic blood pressure (BP) < 80 mmHg or ≥ 150 mmHg, Diastolic BP < 50 mmHg or ≥ 95 mmHg, Pulse < 50 bpm or > 100 bpm, Signs of pulmonary oedema or volume overload, Any clinically significant rhythm, conduction, or morphology abnormalities in the ECG including but not limited to QT interval corrected using Fridericia's formula (QTcF) > 450 ms.

For female participants only - currently pregnant (confirmed with positive pregnancy test) or breastfeeding.

* Current smokers or participants with smoking history ≥ 10 pack-years.
* Participants with a known long-term exposure to occupational asbestos, silica, radon, heavy metals, and polycyclic aromatic hydrocarbons.
* Positive, first-degree family history of primary lung cancer.
* Positive urine cotinine test at Visit 1 and at any timepoint throughout the study.
* Major surgery within 8 weeks prior to Visit 1, or planned inpatient surgery, major dental procedure or hospitalisation during screening, treatment, or follow-up periods.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2024-08-05 (Actual); Primary Completion 2025-10-15 (Actual); Study Completion 2025-10-15 (Actual)

PRIMARY OUTCOMES:
Change from baseline to end of investigational medicinal product (IMP) administration in expression of T2 and non-T2, and JAK1-related genes and gene signatures in bronchial brushings | 4 weeks
  Gene expression in airway epithelial cells

SECONDARY OUTCOMES:
Change from baseline to end of IMP administration in STAT phosphorylation in bronchial biopsies | 4 weeks
  To evaluate the effect of AZD4604 as compared to placebo on STAT phosphorylation in the airways
Change in number of airway cells, including but not limited to inflammatory cells, airway smooth muscle cells, and goblet cells from baseline to end of IMP administration in bronchial biopsies (cells per mm² determined by microscopic evaluation) | 4 weeks
  To explore the effect of AZD4604 on cellular pathology in the airways as compared to placebo

CONTACTS AND LOCATIONS:
Locations (18):
- Canada (4):
  - Research Site, Calgary, Alberta
  - Research Site, Vancouver, British Columbia
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
- Research Site, København NV, Denmark
- Germany (2):
  - Research Site, Frankfurt
  - Research Site, Großhansdorf
- Spain (3):
  - Research Site, Barcelona
  - Research Site, Palma de Mallorca
  - Research Site, Santander
- United Kingdom (8):
  - Research Site, Birmingham
  - Research Site, Glasgow
  - Research Site, Headington
  - Research Site, Leicester
  - Research Site, Liverpool
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Southampton

REFERENCES:
- [Derived] Dosanjh DPS, Darrah E, Jensen TJ, Jevnikar Z, Halvorson A, Cardner M, Hughes R, Grant SS, Platt A, Brightling CE. ARTEMISIA: a mechanistic study of a novel Janus kinase 1 inhibitor to advance molecular understanding and precision medicine in asthma. Respir Res. 2025 Jul 2;26(1):233. doi: 10.1186/s12931-025-03309-3. PMID 40604958